CLINICAL TRIAL: NCT05038332
Title: A Phase II Randomized Trial of Moderate Versus Ultra-hypofractionated Post-prostatectomy Radiation Therapy
Brief Title: Post-prostatectomy Radiation Therapy--Moderate Versus Ultra-hypofractionated (Also Known as Stereotactic Body Radiation Therapy [SBRT])
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: University of Michigan Rogel Cancer Center (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: UMCC 2021.046; HUM00200905 (Other: University of Michigan)
Record Dates: First submitted 2021-08-31; First posted 2021-09-09 (Actual); Last update posted 2026-01-16 (Actual); Status verified 2026-01

CONDITIONS: Prostate Cancer
Keywords: Stereotactic Body Radiation Therapy (SBRT); Ultra-hypofractionated Radiation Therapy; Post-prostatectomy
MeSH Terms: conditions — Prostatic Neoplasms | interventions — Radiosurgery

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: Yes

ARMS (2):
- Moderately Hypo-fractionated Radiation Therapy (Active Comparator): 20 fractions of moderately hypofractionated radiation therapy over no more than 5-6 weeks.
  Interventions: Radiation: Moderately Hypo-fractionated Radiation Therapy
- Ultra-Hypofractionated Radiation Therapy (Experimental): 5 fractions of ultra-hypofractionated radiation therapy with at least one day between each treatment over the course of no more than 3-4 weeks
  Interventions: Radiation: Ultra-hypofractionated radiation therapy

INTERVENTIONS:
Radiation: Ultra-hypofractionated radiation therapy — 34 Gy in 5 fractions to prostate bed, every other day, M-F, ~2 weeks (25 Gy in 5 fractions to pelvic lymph nodes if included)
  Other Names: stereotactic body radiation therapy [SBRT]
  Arms: Ultra-Hypofractionated Radiation Therapy
Radiation: Moderately Hypo-fractionated Radiation Therapy — 55 Gy in 20 fractions to prostate bed, daily, M-F, 4 weeks (42 Gy in 20 fractions to pelvic lymph nodes if included)
  Arms: Moderately Hypo-fractionated Radiation Therapy

SUMMARY:
The primary purpose of this study is to compare the quality of life (QOL) reported by prostate cancer patients 2 years after treatment with ultra-hypofractionated post-prostatectomy radiation therapy (also known as stereotactic body radiation therapy [SBRT]) versus the self-reported QOL of those treated with moderately hypo-fractionated post-prostatectomy radiation (a current standard of care option).

DETAILED DESCRIPTION:
Conventional or moderately hypo-fractionated radiation therapy are the current standard of care treatment options for men receiving post-prostatectomy radiation therapy. These treatment regimens typically span 4-8 weeks, representing a high burden of therapy, which may result in decreased utilization of salvage radiotherapy, the only potentially curable treatment for men with relapsed disease following prostatectomy. Ultra-hypofractionated radiation therapy (also known as stereotactic body radiation therapy [SBRT]) would decrease the total number of treatments to 5, delivered over 2 weeks, which would greatly reduce treatment burden.

ELIGIBILITY:
Inclusion Criteria:

* Men age ≥ 18 with histologically confirmed prostate cancer after radical prostatectomy with a PSA ≥ 0.1 ng/mL
* Interval between prostatectomy and planned radiation therapy start date ≥ 6 months
* KPS ≥ 70
* Patients with equivocal pelvic lymph nodes on imaging are eligible if the nodes are ≤ 1.5 cm in the short axis (equivocal evidence of metastatic disease outside of the pelvis on standard imaging requires documented negative biopsy)
* Ability to complete the EPIC-26 quality of life questionnaire
* Ability to obtain tissue from radical prostatectomy specimen for review by Michigan Medicine Pathology
* Ability to understand and the willingness to sign a written informed consent.

Exclusion Criteria:

* Prior history of pelvic radiation therapy
* History of moderate/severe or active Crohn's disease or ulcerative colitis
* History of bladder neck or urethral stricture
* Evidence of distant metastatic disease or nodal involvement beyond the common iliac vessels
* Initiation of androgen deprivation therapy with a LHRH / GnRH agonist or antagonist greater than 6 months prior to enrollment or receipt of any non-LHRH / GnRH agonist or antagonist androgen deprivation or anti-androgen therapy
* History of another invasive malignancy within the previous 3 years except for adequately treated squamous or basal cell skin cancer
* Any condition that in the opinion of the investigator would preclude participation in this study

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 136 (Estimated)
Dates: Start 2021-11-12 (Actual); Primary Completion 2026-11 (Estimated); Study Completion 2029-11 (Estimated)

PRIMARY OUTCOMES:
Change in patient reported GI and GU quality of life (QOL) at 2-years post-treatment from baseline | 2-years post-treatment
  GI and GU QOL assessed with the EPIC-26 questionnaire, bowel and urinary domains. Change scores will be calculated as baseline score subtracted from 2-year score. All patients with EPIC bowel and urinary domain scores will be included in the primary endpoint analysis. The EPIC scoring manual will be followed which requires ≥ 80% of items in a domain to be completed in order to obtain a score for that domain. High bowel score >96, low bowel score <= 96, high urinary score > 84, low urinary score <=84.

SECONDARY OUTCOMES:
Patient reported GU quality of life (QOL) up to 60 months | 60 months post-treatment
  GU QOL assessed with the EPIC-26 questionnaire, urinary domain; at the end of radiation, 3, 6, 12, and 60 months post-treatment. The EPIC scoring manual will be followed which requires ≥ 80% of items in a domain to be completed in order to obtain a score for that domain. High urinary score > 84, low urinary score <=84. A longitudinal analysis incorporating all follow-up time points, will be conducted separately for each domain score.
Patient reported GI quality of life (QOL) up to 60 months | 60 months post-treatment
  GI QOL assessed with the EPIC-26 questionnaire, bowel domain; at the end of radiation, 3, 6, 12, and 60 months post-treatment. The EPIC scoring manual will be followed which requires ≥ 80% of items in a domain to be completed in order to obtain a score for that domain. High bowel score >96, low bowel score <= 96. A longitudinal analysis incorporating all follow-up time points, will be conducted separately for each domain score.
Treatment related toxicity - acute | ≤ 90 days after treatment completion
  Treatment related toxicity (adverse events) assessed with CTCAE version 5.0
Treatment related toxicity - late | >90 days after treatment completion, up to 5 years
  Treatment related toxicity (adverse events) assessed with CTCAE version 5.0
Time to progression | up to 5 years
  Time to progression (where progression is defined as the first occurrence of biochemical failure, local failure, regional failure, distant metastasis, start of salvage therapy, or death from prostate cancer)
Rate of biochemical failure | up to 5 years
  Biochemical failure will be assessed using two definitions. Definition one is a PSA ≥ 0.4 ng/mL followed by a second higher value. Definition two is the post-radiation PSA nadir + 2ng/mL
Local failure, Regional failure, Distant metastases | up to 5 years
  Descriptive statistics will be used to describe the number of local, regional and distant metastases.
  * Local failure is defined as development of a new biopsy-proven mass or prostate specific PET avid mass in the prostate bed after completion of protocol treatment
  * Regional failure is defined as radiographic evidence of pelvic lymphadenopathy (lymph node size ≥ 1.5 cm in short axis) or PET avid lymph nodes within the pelvis following protocol treatment
  * Distant metastases is defined as any clinical or radiographic evidence of lymph node, bone, or visceral involvement of prostate cancer
Prostate cancer specific survival | up to 5 years
  Prostate cancer specific survival defined as the duration of time from the start of treatment to death attributable to prostate cancer. Patients who have not died or die of non-prostate cancer related causes will be censored at the date of last known follow-up or date of death, respectively.
Overall survival | up to 5 years
  Overall survival defined as the duration of time from the start of treatment to death from any cause. Patients who have not died will be censored at the date of last known follow-up.

CONTACTS AND LOCATIONS:
Overall Officials: William Jackson, M.D., Principal Investigator — University of Michigan Rogel Cancer Center
Locations (1):
- University of Michigan Rogel Cancer Center, Ann Arbor, Michigan, United States

IPD SHARING:
Plan to Share IPD: No